CLINICAL TRIAL: NCT06143176
Title: Efficacy of Virtual Reality in Upper Extremity Rehabilitation for Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, MinYoung Kim, MD, PhD, Principle investigator, Bundang CHA Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-08-032
Record Dates: First submitted 2023-11-13; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Control group will be recruited by propensity matching with the experimental group according to the dataset from retrospective data
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stroke patients (Experimental)
  Interventions: Behavioral: VR-based occupational therapy

INTERVENTIONS:
Behavioral: VR-based occupational therapy — All patients will undergo 20 sessions of virtual reality based occupational therapy for 30 minutes a day, 5 days a week for 4weeks

SUMMARY:
To investigate the therapeutic effect of including virtual reality-based digital content in the upper limb motor function rehabilitation of stroke patients and to develop a treatment method to improve the upper limb motor function of stroke patients in the future.

ELIGIBILITY:
1. Inclusion Criteria for experimental group:

1. Patients aged 19 to 80 years with unilateral stroke within 6 months of stroke onset
2. Motor function evaluation: Patients showing moderate or lower upper limb dysfunction with an upper limb FMA (Fugl-Meyer Assessment) score of less than 58 points on the affected side.
3. Patients receiving or planning to receive exercise rehabilitation treatment 5 days a week

2. Inclusion Criteria for control group:

1) Patients who have been admitted to our hospital's rehabilitation medicine department and received rehabilitation treatment within the past 5 years 2) Patients with unilateral stroke within 6 months of stroke onset who are between 19 and 80 years old at the time of hospitalization 3) Patients who were admitted to the rehabilitation medicine department of our hospital and received exercise rehabilitation treatment for 4 weeks, 5 days a week 4) Patients with similar characteristics below compared to the test group

* Age: Difference within 5 years
* Gait function: Functional Ambulatory Category (FAC)
* Upper extremity function: Fugl-Meyer Assessment (FMA) difference within 6 points
* Cognitive function: Korean Version of Mini Mental State Examination (K-MMSE) difference within 5 points
* Daily living skills: Korean Version of Modified Barthel Index (K-MBI) difference within 10 points

  3. Exclusion Criteria:
  1. Accompanying existing serious neurogenic disease
  2. Cases accompanied by existing serious psychiatric diseases such as major schizophrenia, bipolar disorder, dementia, etc.
  3. Cases where it is difficult to understand task performance due to severe cognitive decline (Korean Mini-Mental State Examination, K-MMSE 10 points or less)
  4. If there are difficulties in conducting research
  5. Other patients who are judged by the principal investigator to have difficulty participating in this study.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-11-27 (Estimated); Primary Completion 2024-11-27 (Estimated); Study Completion 2024-11-27 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment of upper extremity | baseline, 4 weeks after intervention
  Fugl-Meyer assessment for motor function of upper extremity in score

SECONDARY OUTCOMES:
Korean version of modified Barthel index | baseline, 4 weeks after intervention
  Korean version of modified Barthel index for functional status in score
Korean version of mini mental state examination | baseline, 4 weeks after intervention
  Korean version of mini mental state examination for cognitive function in score
Grip and pinch strength test | baseline, 4 weeks after intervention
  Grip and pinch strength test for hand and finger strength in score
Nine-hole pegboard test | baseline, 4 weeks after intervention
  Nine-hole pegboard test for dexterity in seconds
Motion analysis | baseline, 4 weeks after intervention
  Motion analysis is a process of measuring and evaluating kinematic and kinetic parameters including moment (Nm/kg) and power(Nm/s*Kg) of each joint through Qualisys motion analysis system

IPD SHARING:
Plan to Share IPD: No